CLINICAL TRIAL: NCT04475367
Title: Evaluation of the Effect of an APP in Improving Treatment Adherence in Hypertensive Patients in Hypertension Ambulatory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Paula Reis, Nurse Specialist, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 5701-19
Record Dates: First submitted 2020-05-29; First posted 2020-07-17 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Blood Pressure; Adhesion
Keywords: software; hypertension; technology
MeSH Terms: conditions — Tissue Adhesions; Hypertension

STUDY DESIGN:
Intervention Model Description: The participants will be randomized into 2 intervention groups
Who Masked: Outcomes Assessor
Masking Description: blind research assistant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypertensive patients using HyperCrossApp (Experimental): Interdisciplinary health care
  + HyperCross App
  Interventions: Other: App hypercross group
- hypertensive patients without using HyperCrossApp (Active Comparator): Interdisciplinary health care
  Interventions: Other: without App hypercross group

INTERVENTIONS:
Other: App hypercross group — hypertensive patients using HyperCrossApp
  Arms: hypertensive patients using HyperCrossApp
Other: without App hypercross group — Interdisciplinary health care
  Arms: hypertensive patients without using HyperCrossApp

SUMMARY:
Brief Summary: Through the App, the user will have the opportunity to connect directly with the health professional, clarify doubts and manage the treatment of their hypertension.

DETAILED DESCRIPTION:
To evaluate treatment adherence and blood pressure reduction, through the HiperCross App, between two groups of hypertensive patients in a Hypertension Public Ambulatory in Porto Alegre.

The investigators hope to identify better adherence to treatment, as well as a significant reduction in blood pressure, all of these results will be better evaluated using the HiperCross application.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive patients admitted to the hypertension clinic at Instituto de Cardiologia
* older 18 years

Exclusion Criteria:

* Patients without a mobile phone compatible with the App

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-07-10 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure value | 15 minutes
  systolic Blood pressure and dyastolic Blood pressure

SECONDARY OUTCOMES:
Morisky scale | 15 minutes
  Medication adherence. The Morisky scale condition and medication specific assessment: 1) measures the level of adherence an medication, 2) measures the severity of Major Depressive Disorder, a determinant of non-adherence 3) identifies why the patient is not taking their medication, 4) determines the risk between non-adherence to BP measures of disease control. 0-1 = Low motivation; 2-3 = High motivation / 0-1 = Low knowledge; 2-3 = High knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Eibel, PhD, Study Director — Post Graduation professor - Cardiology Foundation